CLINICAL TRIAL: NCT02200653
Title: A Prospective, Randomised, Double-Blind, Double-Dummy, Titration-to-Response Trial Comparing MICARDIS® (Telmisartan) (40 or 80 mg p.o. Once Daily) and COZAAR® / LORZAAR® (Losartan) (50 or 100 mg p.o. Once Daily) in Patients With Mild-to-Moderate Hypertension Using Ambulatory Blood Pressure Monitoring (TOPAS STUDY = Telmisartan and LOsartan ComParative ABPM Study)
Brief Title: A Trial Comparing MICARDIS® (Telmisartan) and COZAAR® / LORZAAR® (Losartan) in Patients With Mild-to-Moderate Hypertension Using Ambulatory Blood Pressure Monitoring (ABPM)
Acronym: TOPAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.344
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Losartan

ARMS (4):
- Low dose of MICARDIS® (Experimental)
  Interventions: Drug: Low dose of MICARDIS®, once daily; Drug: Placebo
- High dose of MICARDIS® (Experimental)
  Interventions: Drug: High dose of MICARDIS®, once daily; Drug: Placebo
- Low dose of COZAAR® / LORZAAR® (Active Comparator)
  Interventions: Drug: Low dose of COZAAR® / LORZAAR®, once daily; Drug: Placebo
- High dose of COZAAR® / LORZAAR® (Active Comparator)
  Interventions: Drug: High dose of COZAAR® / LORZAAR®, once daily; Drug: Placebo

INTERVENTIONS:
Drug: High dose of MICARDIS®, once daily
  Other Names: Telmisartan
  Arms: High dose of MICARDIS®
Drug: Low dose of MICARDIS®, once daily
  Other Names: Telmisartan
  Arms: Low dose of MICARDIS®
Drug: Low dose of COZAAR® / LORZAAR®, once daily
  Other Names: Losartan
  Arms: Low dose of COZAAR® / LORZAAR®
Drug: High dose of COZAAR® / LORZAAR®, once daily
  Other Names: Losartan
  Arms: High dose of COZAAR® / LORZAAR®
Drug: Placebo

SUMMARY:
The primary aim of the trial is to compare the influence of MICARDIS® (telmisartan) and COZAAR® / LORZAAR® (losartan) in lowering ambulatory diastolic blood pressure (DBP) during the last 6 hours of the 24-hour dosing interval as measured by ABPM. Secondary objectives include evaluations of: 1) change from baseline in mean systolic blood pressure (SBP) during the last 6 hours of the 24-hour dosing interval as measured by ABPM, 2) changes from baseline in SBP and DBP during other periods during the 24-hour ABPM profile, 3) changes from baseline in mean seated trough SBP and DBP as measured by manual cuff sphygmomanometer, and 4) responder rates based on both ABPM and trough cuff blood pressure

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-moderate hypertension defined as a mean seated diastolic blood pressure of ≥ 95 mmHg and ≤ 109 mmHg, measured by manual cuff sphygmomanometer, at Visit 3 (baseline cuff BP)
* A 24-mean DBP of ≥ 85 mmHg at Visit 4 as measured by ABPM
* Age 18 years or older
* Ability to stop current antihypertensive therapy without risk to the patient (investigator's discretion)
* Patient's written informed consent in accordance with good clinical practice (GCP) and local legislation

Exclusion Criteria:

* Pre-menopausal women (last menstruation ≤ 1 year prior to start of run-in period) who:

  * are not surgically sterile; and/or
  * are nursing
  * are of child-bearing potential and are NOT practising acceptable means of birth control, do NOT plan to continue using this method throughout the study. Acceptable methods of birth control include oral, implantable or injectable contraceptives
* Known or suspected secondary hypertension
* Mean sitting SBP ≥ 180 mmHg or mean sitting DBP ≥ 110 mmHg during any visit of the placebo run-in period
* Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

  * Serum glutamate-pyruvate-transaminase (alanine aminotransferase) or serum glutamate-oxaloacetate-transaminase (aspartate aminotransferase) > than 2 times the upper limit of normal range
  * Serum creatinine > 2.3 mg/dL (or > 203 µmol/l)
* Bilateral renal artery stenosis; renal artery stenosis in a solitary kidney; patients post-renal transplant or with only one kidney
* Clinically relevant sodium depletion, hypokalaemia, or hyperkalaemia
* Uncorrected volume depletion
* Primary aldosteronism
* Hereditary fructose intolerance
* Biliary obstructive disorders
* Patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin II receptor antagonists
* History of drug or alcohol dependency within 6 months
* Chronic administration of any medications known to affect blood pressure, except medications allowed by the protocol
* Any investigational therapy within one month of signing the informed consent form
* Congestive heart failure (NYHA functional class congestive heart failure (CHF) class III-IV)
* Unstable angina within the past six months
* Stroke within the past six months
* Myocardial infarction or cardiac surgery within the past six months
* Percutaneous transluminal coronary angioplasty (PTCA) within the past six months
* Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator
* Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve
* Patients with insulin-dependent diabetes mellitus whose diabetes hast not been stable and controlled for at least the past three months as defined by an HbA1c ≥ 10%
* Night shift workers who routinely sleep during the daytime and whose work hours include midnight to 4:00 ante meridiem (AM)
* Known hypersensitivity to any component of the formulations
* Any clinical condition which, in the opinion of the investigator would not allow safe completion of the protocol and safe administration of trial medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2000-05; Primary Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean diastolic blood pressure | Up to 8 weeks after start of treatment
  Measured during the last 6 hours of the 24-hour dosing interval using ABPM

SECONDARY OUTCOMES:
Change from baseline in mean systolic blood pressure | Up to 8 weeks after start of treatment
  Measured during the last 6 hours of the 24-hour dosing interval using ABPM
Changes from baseline in diastolic and systolic blood pressure | Up to 8 weeks after start of treatment
  Measured during other times of the 24-hour ABPM profile (e.g. 24-hour mean, morning mean, daytime mean and nighttime mean)
Changes from baseline in mean seated trough diastolic blood pressure and systolic blood pressure | Up to 8 weeks after start of treatment
  Triplicate measurement in two minute intervals after 5 minutes of rest, in seated position using sphygmomanometer
Assessment of responder rates on ABPM | Baseline, 8 weeks after start of treatment
Assessment of responder rates on trough cuff blood pressure | Baseline up to 8 weeks after start of treatment